CLINICAL TRIAL: NCT06093867
Title: A Prospective Approach for the Early Detection of Infectious and Noninfectious Lung Diseases Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Early Detection of Infectious and Noninfectious Lung Diseases Following Allogeneic Hematopoietic Stem Cell Transplantation
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001742; 001742-H
Record Dates: First submitted 2023-10-20; First posted 2023-10-23 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08-14

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Keywords: allogeneic hematopoietic stem cell transplantation (HSCT); early detection of inflammatory injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- allogeneic HSCT: Up to 30 men or women, 18 - 70 years of age, who are being treated with allogeneic HSCT for a hematologic malignancy, blood, or immune system disorder at the NIH Clinical CenterUp to 10 children 5 - 17 years of age who are being treated with allogeneic HSCT for a hematologic malignancies, blood, or immune system disorder at the NIH Clinical CenterNIH Clinical Center

SUMMARY:
Background:

Stem cell transplants (called hematopoietic stem cell transplantation, or HSCT) are used to treat various diseases. But when the cells for this procedure are donated by someone other than the person who receives the HSCT ( allogeneic HSCT ), the recipient has an increased risk of lung inflammation and scarring. This happens when their immune cells attack healthy lung cells. In this natural history study, researchers will look for the best ways to detect developing lung inflammations earlier after an HSCT.

Objective:

To see if certain tests can detect early signs of lung inflammation in people after HSCT.

Eligibility:

People aged 5 to 70 years who will have HSCT as part of another NIH study.

Design:

Participants will undergo these tests prior to their HSCT. These tests will then be repeated regularly for 2 years:

Ultra-low dose computed tomography (CT) scans. Participants will lie on a table that slides through a machine; the machine uses X-rays to get pictures of the inside of the body. This type of scan uses less radiation than normal CT scans.

Bronchoscopy with lavage: Participants will be sedated. A flexible tube will be inserted through the mouth and into the airways. Salt water will be squirted into the lung, then sucked out to collect cells and fluids from the lung. Another tube with a camera may be inserted into the airways to take pictures.

Blood tests. Blood will be drawn every 2 to 4 weeks.

Pulmonary function tests. Participants will breathe into a machine to test their lung function. They will see how far they can walk in 6 minutes.

DETAILED DESCRIPTION:
Study Description:

The primary goal of this proposal is to use preemptive pulmonary imaging, biomarker measurement with surveillance bronchoscopy to improve the early detection of inflammatory injury after allogeneic hematopoietic stem cell transplantation (HSCT). These data may provide early identification of patients at risk for infectious and noninfectious lung diseases and accelerate the development of targeted therapies.

Objectives:

Primary Objective:

To use preemptive assessments with sequential chest imaging and bronchoalveolar lavage (BAL) measures to provide earlier identification of lung injury due to infection or alloreactive lung syndromes associated with hematopoietic stem cell transplantation

Secondary Objectives:

To use high density proteomic, transcriptomic and metagenomic analysis of specimens from the lung and blood to define mechanisms of altered lung function associated with HSCT.

Endpoints:

Primary Endpoint: To assess whether surveillance chest tomography and bronchoscopy with lavage detects incipient lung infection and noninfectious lung injury prior to and following HSCT

Secondary Endpoints: To determine if biomarkers from surveillance proteomic, transcriptomic or metagenomic analysis will provide early identification of lung injury prior to the development chronic progressive and irreversible lung disease

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Male or female, aged 5 - 70 years of age
3. Are to be treated with allogeneic HSCT for a hematologic malignancy, blood, or immune system disorders at the NIH Clinical Center.
4. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnancy or lactation

a. HSCT is not available to pregnant women or lactating women in the intramural program. For women of reproductive potential, have a negative serum pregnancy test during the screening period. Women of reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion; or who have not been naturally postmenopausal (i.e., who have not menstruated at all for at least the preceding 1 year prior to signing informed consent unrelated to hormonal contraception).

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men or women, 18 - 70 years of age & children 5 - 17 years , who are being treated with allogeneic HSCT for a hematologic malignancy, blood, or immune system disorder at the NIH Clinical Center
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
To use preemptive assessments with sequential chest imaging and BAL measures to provide earlier identification of lung injury due to infection or alloreactive lung syndromes associated with HSCT. | 30 months
  To assess whether surveillance chest tomography and bronchoscopy with lavage detects incipient lung infection and noninfectious lung injury prior to and following HSCT

SECONDARY OUTCOMES:
To use high density proteomic, transcriptomic and metagenomic analysis of specimens from the lung and blood to define mechanisms of altered lung function associated with HSCT. | 30 months
  To determine if biomarkers from surveillance proteomic, transcriptomic or metagenomic analysis will provide early identification of lung injury prior to the development chronic progressive and irreversible lung disease

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F Suffredini, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Refer to the DMSP
Supporting Information: Study Protocol, ICF

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001742-H.html